CLINICAL TRIAL: NCT06610734
Title: Multicenter, Phase II Randomized Controlled Study of Adebrelimab Combined With Chemotherapy and Concurrent Low-Dose Radiotherapy (LDRT) for the Treatment of Extensive-Stage Small Cell Lung Cancer (SCLC)
Acronym: SKY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Collaborators: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, You Lu, Chief of Thoracic Cancer Ward, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKY; 2024 Review (No. 1573) (Other: Biomedical Ethics Review Committee of West China Hospital of Sichuan University)
Record Dates: First submitted 2024-09-14; First posted 2024-09-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: SCLC; Adebrelimab; LDRT
MeSH Terms: interventions — Immunotherapy; Immune Checkpoint Inhibitors; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Adebrelimab combined with chemotherapy synchronous LDRT
  Interventions: Drug: Adebrelimab; Drug: Chemotherapy; Radiation: low dose radiotherapy
- Group B (Active Comparator): Adebrelimab combined with chemotherapy
  Interventions: Drug: Adebrelimab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab combined with chemotherapy synchronous LDRT
  Other Names: immunotherapy; Programmed death ligand 1 inhibitor
Drug: Chemotherapy — Chemotherapy
Radiation: low dose radiotherapy — low dose radiotherapy
  Arms: Group A

SUMMARY:
Multicenter, Phase II Randomized Controlled Study of Adebrelimab Combined with Chemotherapy and Concurrent Low-Dose Radiotherapy (LDRT) for the Treatment of Extensive-Stage Small Cell Lung Cancer (SCLC)

DETAILED DESCRIPTION:
Multicenter, Phase II Randomized Controlled Study of Adebrelimab Combined with Chemotherapy and Concurrent Low-Dose Radiotherapy (LDRT) for the Treatment of Extensive-Stage Small Cell Lung Cancer (SCLC)

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 75 years, regardless of gender;
* ECOG Performance Status (PS) score of 0-1;
* Expected survival duration of no less than 8 weeks;
* Histologically or cytologically confirmed extensive small cell lung cancer (according to the VALG staging system);
* Subjects must not have received systemic therapy or radical radiotherapy for extensive SCLC prior to enrollment.

Exclusion Criteria:

* Tissue classifications of mixed small cell lung cancer and non-small cell lung cancer;
* Patients who have undergone major surgical procedures within 28 days prior to the initial administration of the study drug, or those planning to undergo major surgery during the study period (as determined by the investigator);
* Receipt of live attenuated vaccines within 28 days before the first dose or planned for the duration of the study;
* Participation in another clinical trial within 28 days preceding initial dosing, involving any experimental agents;
* History of receiving chest radiotherapy or plans for intensive chest radiotherapy prior to systemic therapy;
* Any previous T-cell co-stimulation or immune checkpoint therapies administered;
* Documented history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation."

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | From date of randomization to the time when the subject died from any cause, up to approximately 36 months
  Time from randomization to death from any cause. Unit of measure: median overall survival (months); hazard ratio (HR) and 95% confidence interval (CI); 12- and 24-month survival rates (%).
  Assessment schedule: survival status assessed every 3 months after the end of treatment until death or study cut-off (up to 36 months).

SECONDARY OUTCOMES:
Progression free survival | From date of randomization to the date of documented progression or death from any cause, whichever occurs first, assessed up to 36 months.
  Time from randomization to the earliest of radiologically documented progressive disease (per RECIST 1.1 assessed by the investigator) or death from any cause.
  Unit of measure: median progression-free survival (months); hazard ratio (HR) and 95% confidence interval (CI); 6- and 12-month PFS rate (%).
  Measurement tool: contrast-enhanced CT or MRI scanned every 6 weeks for the first 48 weeks, then every 12 weeks until disease progression, death, or study cut-off.
Time to second progression or death (PFS2) | From date of randomization to the date of second documented progression or death from any cause, whichever occurs first, assessed up to 36 months
  Defined as time from randomization to the earliest of radiologically documented second progression (per RECIST 1.1 assessed by the investigator ) or death from any cause.
  Unit of measure: median PFS2 (months); hazard ratio (HR) and 95% CI; 6- and 12-month PFS2 rate (%).
  Measurement tool: contrast-enhanced CT/MRI. Assessment schedule: imaging every 6 weeks during induction; every 4-6 weeks during maintenance; after first PD, every 6 weeks until second PD or death.
Disease control rate | From date of randomization until disease progression, death, or 24 months, whichever occurs first.
  Proportion of randomized subjects with best overall response of complete response (CR), partial response (PR), or stable disease (SD) per RECIST 1.1 assessed by the investigator.
  Unit of measure: percentage of patients (%); 95% confidence interval (Clopper-Pearson).
  Assessment schedule: scans every 6 weeks for the first 48 weeks, then every 12 weeks until progression, death, or 36 months.
Overall response rate (ORR) | From date of randomization until disease progression, death, or 24 months, whichever occurs first
  Proportion of randomized subjects achieving complete response (CR) or partial response (PR) per RECIST 1.1 assessed by the investigator.
  Unit of measure: percentage of patients (%); 95% confidence interval (Clopper-Pearson).
  Assessment schedule: scans every 6 weeks (±7 days) for the first 48 weeks, then every 12 weeks (±7 days) until progression, death, or 36 months; response determined by site investigator.
Duration of response (DoR) | From the date of first CR/PR to the date of documented progression or death from any cause, assessed up to 36 months
  Time from first documented complete response (CR) or partial response (PR) per RECIST 1.1 (investigator assessment) until the date of documented progressive disease or death from any cause, whichever occurs first.
  Unit of measure: median duration of response (months); 95% confidence interval of the median; 6- and 12-month response duration rate (%) Assessment schedule: imaging every 6 weeks for the first 48 weeks, then every 12 weeks until progression, death, or 36 months.
Depth of Response | From date of randomization until disease progression, death, or 24 months, whichever occurs first.
  Maximum percentage reduction in the sum of longest diameters of target lesions relative to baseline per RECIST 1.1 assessed by the investigator.
  Unit of measure: median percentage change (%); inter-quartile range (IQR); Assessment schedule: scans every 6 weeks for the first 48 weeks, then every 12 weeks until progression, death, or 36 months; tumor diameters measured by the site investigator.
Post-progression survival (PPS) | From the date of documented progression to the date of death from any cause, assessed up to 36 months after progression.
  Time from the date of first documented progressive disease (per RECIST 1.1, investigator assessment) to the date of death from any cause.
  Unit of measure: median post-progression survival (months); hazard ratio (HR) and 95% confidence interval; 6- and 12-month survival rate (%).
  Assessment schedule: survival status contacted every 3 months after progression until death, lost to follow-up, or study cut-off.
Incidence and severity of adverse events (AEs) | Collect and assess safety-related test results and adverse events (AEs) for both the experimental group and the control group during the first-line and second-line treatment phases (to 90 days after the last dose of drug).
  Number and percentage of participants experiencing AEs graded per CTCAE v5.0 by the treating investigator.
  Unit of measure: incidence rate (%); number of events; severity distribution (Grade 1-5).
  Measurement tool: investigator assessment using CTCAE v5.0. Assessment schedule: continuous monitoring from informed consent through 90 days after last dose of study drug; assessed at every study visit (baseline, weekly during cycle 1, then day 1 of each subsequent cycle, and at follow-up).
Incidence of serious adverse events (SAEs) | Collect and assess safety-related test results and adverse events (AEs) for both the experimental group and the control group during the first-line and second-line treatment phases(before 2nd PD and 3 month afterwords).
  Number and percentage of participants experiencing serious adverse events (SAE) graded per CTCAE v5.0 by the treating investigator.
  Unit of measure: incidence rate (%) of subjects with ≥1 SAE; number of events; severity distribution (Grade 1-5).
  Measurement tool: investigator assessment using CTCAE v5.0. Assessment schedule: continuous monitoring from informed consent through 90 days after last dose of study drug. All SAEs reported within 24h of awareness.

OTHER OUTCOMES:
Correlation of PD-L1 expression with overall survival | From baseline to death from any cause, assessed up to 36 months
  Pearson correlation coefficient between baseline PD-L1 expression and overall survival (months).
  Unit of measure: r (dimensionless) with 95% confidence interval. Measurement tool: PD-L1 IHC 22C3 pharmDx assay; PD-L1 tumor proportion score (TPS, %).
  Assessment schedule: baseline diagnostic biopsy and, if clinically feasible, at the time of first and second tumor progression.
Correlation of PD-L1 expression with progression-free survival | From date of randomization to the date of documented progression or death from any cause, whichever occurs first, assessed up to 36 months.
  Pearson correlation coefficient between baseline PD-L1 TPS and PFS (months). Unit of measure: r (dimensionless) with 95% CI. Measurement tool: PD-L1 IHC 22C3 pharmDx assay; TPS (%). Assessment schedule: baseline tumor biopsy.
Correlation of neutrophil count with overall survival | From baseline to death from any cause, assessed up to 36 months
  Pearson correlation coefficient between baseline peripheral blood neutrophil count and overall survival (months).
  Unit of measure: r (dimensionless) with 95% CI. Measurement tool: automated hematology analyzer; absolute neutrophil count (10⁹/L).
Patient-Reported Global Health Status and Quality of Life Score | From baseline (pre-treatment) to disease progression or death or initiation of new anti-tumour therapy, assessed up to 36 months
  Change in patient-reported global health status/quality of life score, as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) global health status/quality of life scale (items 29 and 30).
  Unit of measure: Mean change from baseline in score. Scale Details: The EORTC QLQ-C30 global health status/QoL scale is a 7-point Likert scale ranging from 1 ("Very poor") to 7 ("Excellent"). The raw score is linearly transformed to a 0-100 scale. Higher scores indicate a better quality of life.
Patient-Reported Functioning Scale Scores (Composite of Five Scales) | From baseline (pre-treatment) to disease progression or death or initiation of new anti-tumour therapy; assessed up to 36 months.
  Change in patient-reported functioning, as measured by the five functioning scales of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30): physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning.
  Unit of Measure: Mean change from baseline in score for each scale. Scale Details: Each EORTC QLQ-C30 functioning scale consists of multiple items using a 4-point Likert scale (1="Not at all", 4="Very much"). Raw scores are linearly transformed to a 0-100 scale. For functioning scales, higher scores indicate a better level of functioning.
Patient-Reported Lung Cancer Symptom Scale Scores (Composite of Scales) | From baseline (pre-treatment) to disease progression or death or initiation of new anti-tumour therapy; assessed up to 36 months.
  Change in patient-reported lung cancer symptoms, as measured by the symptom scales and items of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13): dyspnoea, cough, haemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, and pain.
  Unit of Measure: Mean change from baseline in score for each symptom scale/item.
  Scale Details: EORTC QLQ-LC13 scales use a 4-point Likert scale (1="Not at all", 4="Very much"), transformed to a 0-100 scale. For symptom scales, higher scores indicate a greater severity of symptoms/worse outcome.
OS in liver-metastasis subgroup | From date of randomization to death from any cause, assessed up to 36 months
  Treatment effect (adebrelimab + chemotherapy ± LDRT vs control) on overall survival in the pre-specified subgroup defined by baseline liver metastasis (yes vs no).
  Unit of measure: hazard ratio (HR) with 95% confidence interval; median overall survival (months); 12-month survival rate (%).
  Measurement tool: death from any cause determined by medical records or death registry.
OS in brain-metastasis subgroup | From date of randomization to death from any cause, assessed up to 36 months.
  Treatment effect on overall survival in the subgroup defined by baseline brain metastasis (yes vs no).
  Unit of measure: HR with 95% CI; median OS (months); 12-month survival rate (%).
  Measurement tool: death from any cause determined by medical records or death registry.
PFS in liver-metastasis subgroup | From date of randomization to the date of documented progression or death from any cause, whichever occurs first, assessed up to 36 months.
  Treatment effect on PFS (RECIST 1.1, investigator) in the liver-metastasis subgroup (yes vs no).
  Unit of measure: HR with 95% CI; median PFS (months); 6-month PFS rate (%). Measurement tool: CT/MRI.
PFS in brain-metastasis subgroup | From date of randomization to the date of documented progression or death from any cause, whichever occurs first, assessed up to 36 months.
  Treatment effect on PFS in the brain-metastasis subgroup (yes vs no). Unit of measure: HR with 95% CI; median PFS (months); 6-month PFS rate (%). Measurement tool: CT/MRI.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
The survival data of individual participant will be shared after the research is completed.
Supporting Information: Study Protocol, CSR
Time Frame: After the study is completed.
Access Criteria: Other Medical Professionals with permission from Principle Investigator